CLINICAL TRIAL: NCT02765711
Title: TIFU: A Non-Interventional, Descriptive Cohort Study to Describe the Use of Ticagrelor in Patients With Acute Coronary Syndrome (TIFU: Ticagrelor in Fuwai Hospital)
Brief Title: Ticagrelor in Fuwai Hospital
Acronym: TIFU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Hongbing Yan, The deputy director of Center of Coronary Heart Disease and Center of Chest Pain, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016-ZX07; ESR-15-11199 (Other: AstraZeneca)
Record Dates: First submitted 2016-04-24; First posted 2016-05-09 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Acute Coronary Syndrome
Keywords: ticagrelor; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- the use of ticagrelor in hospital

SUMMARY:
This is a single-arm non-interventional cohort study. This study is to describe the contemporary use of ticagrelor in a "real-world" setting, to reflect its acceptance and patients' compliance, and to observe its one-year safety in patients with acute coronary syndrome in Fuwai Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. ≧18 years
2. Established diagnosis of acute coronary syndrome
3. The use of ticagrelor in hospital
4. agree to join this clinical trial and sign informed consent

Exclusion Criteria:

1. Life-expectancy <1 year
2. Dialysis required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include more than 1200 ACS patients using ticagrelor in Fuwai hospital from May 2016 to May 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with switching between clopidogrel and ticagrelor | 12 months
Number of participants with switching between clopidogrel and ticagrelor without a reloading dose | 12 months
Number of Participants with discontinuation of P2Y12 receptor antagonist | 12 months
Number of Participants with ticagrelor combined with other anticoagulants | 12 months

SECONDARY OUTCOMES:
Cardiovascular Mortality, Myocardial Infarction(MI), Ischemic Stoke | 12 months
  composite incidence
  Myocardial infarction is defined and subclassified in accordance with ACC/AHA/ESC third universal definition of myocardial infarction
  Ischemic stroke: an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction, defined by at least one of the following:
  1. Pathological, imaging, or other objective evidence of acute, focal cerebral, spinal, or retinal ischemic injury in a defined vascular distribution
  2. Symptoms of acute cerebral, spinal, or retinal ischemic injury persisting ≧24 h, with other etiologies excluded
  Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke.
Number of bleeding event will be recorded (defined in accordance with PLATO definition) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongbing Yan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China